CLINICAL TRIAL: NCT01922505
Title: The Trend of Eradication Rates of First-line Triple Therapy for Helicobacter Pylori and Clinical Factors That Affect the Eradication in Korean: Single Center Experience for Recent Ten Years
Brief Title: Eradication Rates of Helicobacter Pylori and Its Affecting Factors
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, M.D., Seoul National University Bundang Hospital
Other Study IDs: B-1308-214-108; 2012R1A1A3A04002680 (Other: National Research Foundation of Korea)
Record Dates: First submitted 2013-08-11; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Helicobacter Infections
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PPI triple therapy: 7-day PPI triple therapy regimen: PPI (esomeprazole 40 mg or omeprazole 20 mg or lansoprazole 30 mg or pantoprazole 40 mg or rabeprazole 20 mg) plus amoxicillin (1000mg) and clarithromycin (500mg) twice daily for 7 days.
  Interventions: Drug: PPI triple therapy

INTERVENTIONS:
Drug: PPI triple therapy

SUMMARY:
The purpose of this study is to investigate the trend of eradication rates of first-line triple therapy for Helicobacter pylori in recent ten years and clinical factors that affect the eradication in Korean.

DETAILED DESCRIPTION:
A PPI triple regimen combining a proton pump inhibitor(PPI) with two antibiotics (amoxicillin and clarithromycin) is currently considered the gold standard therapy for eradication of H. pylori. However, recently the eradication rate with first-line treatment has a tendency to decrease because of increasing antibiotics resistance. In addition, PPI is mainly metabolized by cytochrome p450 2C19 (CYP2C19) in the liver and several reports have suggested that differences in th CYP2C19 genotype are associated with H. pylori eradication failure. Thus, the first aim of this study is to investigate the trend of eradication rates of first-line triple therapy in recent ten years. And the second aim is to analyze the antibiotics resistance rate for H. pylori by using culture minimal inhibitory concentrations(MICs) result and to analyze the association between CYP2C19 genotype and eradication rate of H.pylori. And also investigate the other clinical factors (age, gender, underlying disease, cigarette smoking and alcohol use) that affect the eradication rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who proven H. pylori infection by invasive or non-invasive H. pylori test
* Patients treated with First-line triple therapy (PPI + Amoxicillin + Clarithromycin)

Exclusion Criteria:

* Previous eradication therapy for H. pylori
* Follow-up loss patients after eradication therapy
* Other treatment regimen
* Poor medication compliance (<80%)

Ages: 16 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: H. pylori positive patient
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2003-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Eradication Rates of First-line Triple Therapy for Helicobacter pylori | Four weeks after completing eradication therapy
  Non invasive H. pylori test (13C-urea breath test(UBT)) or invasive H. pylori test (Giemsa histology, Rapid Urease test) were performed after four weeks after completing eradication therapy.

SECONDARY OUTCOMES:
Clinical Factors that Affect the Eradication | Four weeks after completing eradication therapy
  Main variables are Cytochrome P450 2C19 (CYP2C19) genotype and Antibiotics resistance by H. pylori culture MICs result.
  Other variables are age, gender, underlying disease (hypertension, diabetes, chronic liver, lung, kidney diseases), cigarette smoking and alcohol use.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Bundang-gu, Seongnam, Gyeonggi-do, South Korea